CLINICAL TRIAL: NCT04359914
Title: Biomarker-guided Assessment of Neurocognitive Impairment in Patients With COVID-19 - a Multicenter Case-control Study
Brief Title: Neurocognitive Impairment in Patients With COVID-19
Acronym: NCoV
Status: Completed | Type: Observational
Sponsor: University of Rostock (Other)
Collaborators: Ludwig-Maximilians - University of Munich (Other); University College, London (Other)
Responsible Party: Principal Investigator, Dr. Johannes Ehler, MD, PD Dr. med. Johannes Ehler, MD, University of Rostock
Other Study IDs: COVID-BRAIN
Record Dates: First submitted 2020-04-19; First posted 2020-04-24 (Actual); Last update posted 2024-01-29 (Actual); Status verified 2024-01

CONDITIONS: Critical Illness; COVID-19; Central Nervous System Injury; Delirium; Encephalopathy
MeSH Terms: conditions — Critical Illness; COVID-19; Delirium; Brain Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- NCoV-A-COVID: * adult patients of every age
  * admission to hospital with suspected COVID-19 disease
  * confirmed SARS-CoV-2 infection within 48 hours after admission
- NCoV-A-CONTROL: * adult patients of every age
  * admission to hospital with suspected COVID-19 disease
  * exclusion of SARS-CoV-2 infection within 48 hours after admission
- NCoV-P-COVID: * pediatric patients
  * admission to hospital with suspected COVID-19 disease
  * confirmed SARS-CoV-2 infection within 48 hours after admission
- NCoV-P-CONTROL: * pediatric patient
  * admission to hospital with suspected COVID-19 disease
  * exclusion of SARS-CoV-2 infection within 48 hours after admission

SUMMARY:
Delirium and acute neurocognitive impairment are increasingly observed in adult and pediatric patients with COVID-19. Prospective clinical studies combining clinical and laboratory examinations including specific biomarkers of neuroaxonal injury were not performed for COVID-19. The value of biomarkers of neuroaxonal injury was proven in preliminary studies. These biomarkers could thus contribute to the systematic detection of neurocognitive impairment in patients with COVID-19. Due to worldwide increasing numbers of hospitalized patients with COVID-19, biomarkers of neuroaxonal injury are highly valuable to detect and monitor cognitive impairment, especially with regard to limited resources available to perform time-consuming brain imaging.

Biomarkers of neuroaxonal injury are therefore not only of great interest to detect neurocognitive impairment but also to quantify the severity of brain injury in patients with COVID-19.

DETAILED DESCRIPTION:
This is a multicenter observational study evaluating the incidence and severity of neurocognitive impairment in adult and pediatric patients with COVID-19. All study participants will be assessed by clinical and neurological examination as well as comprehensive laboratory tests using biomarkers of neuroaxonal injury at study day 1 (day of study inclusion), day 3, day 7 and day of hospital discharge. A panel of biomarkers (among others NSE, S100B and neurofilament proteins) will be measured. Clinical assessment will be performed using validated delirium tests (among others CAM-ICU, ICDSC) and scales to assess the neurocognitive performance of study participants before and three months after study inclusion (among others Short Blessed Test).

A group of patients with a comparable severity of disease but without the detection of SARS-Cov-2 will serve as control group and will undergo the same clinical and laboratory examinations.

We hypothesize, that:

* patients with COVID-19 are more likely to develop delirium and neurocognitive impairment than patients without COVID-19
* patients with a preexisting neurocognitive deficit are more vulnerable to neurocognitive impairment in the course of COVID-19 than patients without a preexisting neurocognitive deficit
* Specific biomarkers of neuroaxonal injury correlate with the clinical severity of acute neurocognitive impairment and can predict the 3-month neurocognitive outcome of patients with COVID-19

ELIGIBILITY:
Inclusion Criteria:

* adult patients of every age
* admission to hospital with suspected COVID-19 disease
* confirmed SARS-CoV-2 infection within 48 hours after admission

Exclusion Criteria:

* transferral from another hospital
* other acute central nervous system diseases (e.g. meningoencephalitis, intracerebral ischemia or hemorrhage)
* confirmed SARS-CoV-2 infection later than 48 hours after hospital admission
* participation in another interventional study
* no written informed consent from patient or legal representative

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with suspected SARS-CoV-2 infection who are admitted to the study centers will be screened for study eligibility according to the inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 118 (Actual)
Dates: Start 2020-04-15 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Incidence of delirium/neurocognitive impairment in adult and pediatric patients with COVID-19 compared to patients without COVID-19 | Day 90
  Assessment of neurocognitive impairment using validated tools
Change in neuroaxonal injury biomarker levels in patients with COVID-19 compared to patients without COVID-19 | Change from baseline biomarker levels at day 28
  Measurement of biomarker levels (e.g. NSE, S100B, neurofilament proteins) derived from blood samples
Neurocognitive 3-months outcome in patients with COVID-19 compared to patients without COVID-19 | Day 90
  Assessment of the neurocognitive performance of patients using validated tests (e.g. Short Blessed Test)
Neurocognitive 3-months outcome in patients with COVID-19 compared to patients without COVID-19 | Change from baseline IQCODE results at day 90
  Assessment of the change in the neurocognitive performance of patients using validated tests (e.g. IQCODE)

SECONDARY OUTCOMES:
Quality of life in patients with COVID-19 compared to patients without COVID-19 after hospital discharge | Day 90
  Assessment of the overall quality of life using validated tests [e.g. Modified Rankin Scale with a range from 0 (no symptoms) to 6 (dead)]
Length of hospital stay in patients with COVID-19 compared to patients without COVID-19 | 1 year
  Cumulative days in hospital
90-day survival in patients with COVID-19 compared to patients without COVID-19 | Day 90
  Survival after 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Ehler, MD, Principal Investigator — University of Rostock
Locations (1):
- Department of Anesthesiology and Intensive Care Medicine, University Medical Center Rostock, Rostock, Mecklenburg-Vorpommern, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ehler J, Klawitter F, von Mollendorff F, Zacharias M, Fischer DC, Danckert L, Bajorat R, Hackenberg J, Bertsche A, Loebermann M, Geerdes-Fenge H, Fleischmann R, Klinkmann G, Schramm P, Schober S, Petzold A, Perneczky R, Saller T. No substantial neurocognitive impact of COVID-19 across ages and disease severity: a multicenter biomarker study of SARS-CoV-2 positive and negative adult and pediatric patients with acute respiratory tract infections. Infection. 2025 Apr;53(2):593-605. doi: 10.1007/s15010-024-02406-7. Epub 2024 Oct 1. PMID 39352661